CLINICAL TRIAL: NCT04586296
Title: Tele-monitoring of Post Join Arthroplasty Outcomes: A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Sameer Naranje, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-300005894
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Post-Op Complication
Keywords: telemedicine; knee replacement; hip replacement
MeSH Terms: conditions — Postoperative Complications | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine Group (Experimental): Group that will be receiving the telemedicine intervention in addition to the standard of care post-op.
  Interventions: Other: Telemedicine
- Standard Treatment (No Intervention): Patients will be receiving the standard of care, post op visits at 2, 6, and 12 weeks.

INTERVENTIONS:
Other: Telemedicine — IVR will consist of a 3 minute call at a decreasing interval from the time of surgery. Questions will assess pain control, signs of infection, prosthesis failure.
  Other Names: Integrated Voice Response (IVR)
  Arms: Telemedicine Group

SUMMARY:
The purpose of this study is to develop an effective telephone mediated follow-up system to reduce the number of unplanned readmissions and emergency department visits after total joint arthroplasty. This will help reduce costs related to unnecessary visits to the hospital as well as catch complications earlier on. The investigators plan to accomplish this by performing a pilot study that will compare the outcomes of using an Interactive Voice Response system through phone call in addition to the standard follow-up protocol. The outcomes of this group will be compared to those receiving the standard of care follow-up protocol.

DETAILED DESCRIPTION:
Upon patient education and consent to participate in this study, patients will be randomized via online randomizer during their baseline visit into either Treatment As Usual (TAU) or Integrated Voice Response (IVR) cohorts. During this baseline visit, the patients in the IVR group will be given specific information on the nature of the calls and what to expect. Both groups will fill out a form for assessing their baseline pain and functionality. Both groups will receive standard total joint arthroplasty. After this, the TAU group will receive the standard of care which involves appropriate pain management and scheduled clinic follow-ups lasting approximately 60 minutes at 2 weeks, 6 weeks, and 12 weeks along with additional visits if required. Clinic visits will assess pain via VAS scale, joint functionality via HOOS and KOOS scale, and quality of life via SF-36.

In addition to the standard of care follow-up visits as in the TAU group, the IVR group will also receive automated phone calls lasting up to 3 minutes, which will be the focus of this research study. These phone calls will be daily for the first week, every other day the second week, twice a week for weeks 3-6, and weekly for weeks 7-12. The content of these calls will assess pain management, wound healing and screen for potential complications through a series of questions (questionnaire script attached). At the completion of each call, the patient will be instructed to either continue standard treatment or visit the emergency department based on the content of their response. If there is reason for concern, the PI will automatically be informed.

Survey questions pertaining to the patients outcomes and satisfaction will be completed in clinic and collected by the PI. The responses and data relating to IVR calls will made available through computer software designed by our team on the secure REDcap network.

ELIGIBILITY:
Inclusion Criteria:

* Participants eligible to undergo the TJA surgical procedure

Exclusion Criteria:

* Participants who are not eligible to undergo the TJA surgical procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-16 (Actual)

PRIMARY OUTCOMES:
Percentage of Patients with acceptable pain control as measured by Visual Analogue scale | 2 week
  VAS is a patient measured scale to evaluate pain, on a scale of 1-10 with 10 being the worst pain.
Percentage of Patients with acceptable pain control as measured by Visual Analogue scale | 6 weeks
  VAS is a patient measured scale to evaluate pain, on a scale of 1-10 with 10 being the worst pain.
Percentage of Patients with acceptable pain control as measured by Visual Analogue scale | 12 weeks
  VAS is a patient measured scale to evaluate pain, on a scale of 1-10 with 10 being the worst pain.
Percentage of Patients with acceptable pain control as measured by Visual Analogue scale | Baseline
  VAS is a patient measured scale to evaluate pain, on a scale of 1-10 with 10 being the worst pain.
Percentage of Patients with acceptable joint functionality as measured by hip disability and osteoarthritis outcome score (HOOS) | Baseline
  HOOS is patient measured scores evaluating Hip function and creates a score out of 100, 100 indicating full functionality.
Percentage of Patients with acceptable joint functionality as measured by hip disability and osteoarthritis outcome score (HOOS) and knee disability and osteoarthritis outcome score (KOOS) | Baseline
  KOOS is a patient measured score evaluating Hip function and creates a score out of 100, 100 indicating full functionality.
Percentage of Patients with acceptable joint functionality as measured by knee disability and osteoarthritis outcome score (KOOS) | 2 weeks
  KOOS is a patient measured score evaluating knee function and creates a score out of 100, 100 indicating full functionality.
Percentage of Patients with acceptable joint functionality as measured by hip disability and osteoarthritis outcome score (HOOS) | 2 weeks
  HOOS is a patient measured score evaluating knee function and creates a score out of 100, 100 indicating full functionality.
Percentage of Patients with acceptable joint functionality as measured by hip disability and osteoarthritis outcome score (HOOS) | 6 weeks
  HOOS is a patient measured score evaluating Hip function and creates a score out of 100, 100 indicating full functionality.
Percentage of Patients with acceptable joint functionality as measured by knee disability and osteoarthritis outcome score (KOOS) | 6 weeks
  KOOS is a patient measured score evaluating knee function and creates a score out of 100, 100 indicating full functionality.
Percentage of Patients with acceptable joint functionality as measured by hip disability and osteoarthritis outcome score (HOOS) | 12 weeks
  HOOS is a patient measured scores evaluating Hip function and creates a score out of 100, 100 indicating full functionality.
Percentage of Patients with acceptable joint functionality as measured by knee disability and osteoarthritis outcome score (KOOS) | 12 weeks
  KOOS is a patient measured score evaluating Hip and knee function and creates a score out of 100, 100 indicating full functionality.
Percentage of Patients with acceptable quality of life as measured by Short Form Health Survey SF-36 | Baseline
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Percentage of Patients with acceptable quality of life as measured by Short Form Health Survey SF-36 | 2 weeks
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Percentage of Patients with acceptable quality of life as measured by Short Form Health Survey SF-36 | 6 weeks
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Percentage of Patients with acceptable quality of life as measured by Short Form Health Survey SF-36 | 12 weeks
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.

CONTACTS AND LOCATIONS:
Overall Officials: Sameer Naranje, MD, Principal Investigator — Assistant Professor
Locations (1):
- UAB Highland Hospital, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No